CLINICAL TRIAL: NCT04580537
Title: Assessing the Efficacy of Image-guided Laser-assisted Enstilar® Delivery for Treatment of Psoriatic Nails - a Proof-of-concept, Single-center, Prospective, Open-label, Randomized, Clinical Trial With an Intra-individual Comparison of Treatments
Brief Title: Assessing the Efficacy of Image-guided Laser-assisted Enstilar® Delivery for Treatment of Psoriatic Nails
Acronym: LAsED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: LEO Innovation Lab (Unknown)
Responsible Party: Principal Investigator, Merete Haedersdal, Sponsor-Investigator [Consultant in dermatology, Clinical professor], Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAsED; 2019-002960-29 (EudraCT Number); H-19047222 (Registry Identifier: De Videnskabsetiske Komitéer)
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Nail Psoriasis
Keywords: Nail disease; Psoriasis; Laser-assisted drug delivery; Enstilar
MeSH Terms: conditions — Nail Diseases; Psoriasis | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Intervention Model Description: a proof-of-concept, single-center, prospective, open-label, randomized, clinical trial with an intra-individual comparison of treatments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser-assisted Enstilar delivery (Experimental): Ablative fractional laser (AFL) pre-treatment + daily use of Enstilar (cutaneous foam: 0.5 mg/g betamethasone dipropionate, 0.05mg/g calcipotriol)
  Interventions: Drug: Enstilar; Device: Ablative fractional laser
- Enstilar (Active Comparator): Daily use of Enstilar (cutaneous foam: 0.5 mg/g betamethasone dipropionate, 0.05mg/g calcipotriol)
  Interventions: Drug: Enstilar

INTERVENTIONS:
Drug: Enstilar — Daily application on affected fingers (nail plates, nail folds, and surrounding skin)
  Other Names: Cutaneous foam
Device: Ablative fractional laser — Pre-treatment of affected fingers (nail plates, nail folds)
  Other Names: AFL
  Arms: Laser-assisted Enstilar delivery

SUMMARY:
The trial is conducted to investigate the clinical efficacy of a combination product containing calcipotriol and betamethasone formulated as an aerosol foam (Enstilar ©) for the treatment of nail psoriasis in conjunction with physical pre-treatment using a fractionally ablative carbon dioxide laser (AFL). It is hypothesized, based on preclinical data and comparable clinical trials, that laser processing prior to topical administration will lead to increased drug distribution, and thereby increase the efficacy of Enstilar® in treating nail psoriasis.

ELIGIBILITY:
Inclusion criteria

1. Informed consent obtained before any trial-related activities.
2. At least 18 years of age (inclusive)
3. Confirmed diagnosis of psoriatic disease with signs of nail psoriasis on at least 2 digits
4. Minimum nail involvement as assessed by treating physician (N-NAIL score of ≥ 2 for at least two individual nails)

Exclusion criteria

1. Insufficient knowledge of written and spoken Danish.
2. Pregnant and lactating women and women who intend to become pregnant during the trial
3. Pre-existing clinical manifestations of long-term side effects of corticosteroid use including but not limited to skin atrophy or telangiectasias on fingers
4. Presence of any skin condition or coloration (marked suntan, hyperpigmentation, smoking-induced staining, tattoos or body art) that would interfere with the evaluation of the clinical response in the test sites or assessment
5. Any non-psoriatic disease activity within test areas
6. Significant history or current evidence of chronic infectious disease, systemic disorders, or organ dysfunction where the use of Enstilar is contraindicated.
7. Known predisposition for hypertrophic scar formation.
8. Known allergy to any of the components of Enstilar®.
9. Current treatment with systemically or locally acting medications which might counter or influence the trial aim
10. Received any drug as part of a research trial within 30 days prior to initial trial dosing.
11. Artificial nail enhancement or damages associated with it, including (semi-) permanent nail polish e.g. acrylic based gels.
12. Ongoing fungal infections of psoriatic nails
13. Close affiliation with the investigator (e.g. a close relative) or persons working at the respective trial site or the participant is an employee of the sponsor
14. In the opinion of the investigator, the participant is unlikely to comply with the Clinical Trial Protocol (e.g. alcoholism, drug dependency or psychotic state).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of topical delivery of Enstilar® with and without laser pre-treatment to improve nail psoriasis | Day1 : Week 24
  Change from baseline to end of treatment in N-NAIL score per nail for each treatment

SECONDARY OUTCOMES:
Safety profile and local tissue response to laser treatment and Enstilar® application | Day 1 : Week 24
  Number of laser- and Enstilar®- emergent adverse events per subject; change in local tissue response score from baseline to Week 12 and Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD PhD DMSc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark